CLINICAL TRIAL: NCT03744780
Title: A One-Day ACT Workshop for Emotional Eating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 143-0818
Record Dates: First submitted 2018-11-02; First posted 2018-11-16 (Actual); Results first posted 2019-11-14 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-10

CONDITIONS: Emotional Eating; Eating Behavior
MeSH Terms: conditions — Emotional Eating; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: All participants will be assigned to the same intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACT Workshop for Emotional Eating (Experimental): All participants will be assigned to a one-day intervention using Acceptance and Commitment Therapy (ACT) techniques to help reduce emotional eating.
  Interventions: Behavioral: ACT Workshop for Emotional Eating

INTERVENTIONS:
Behavioral: ACT Workshop for Emotional Eating — This is a one-day intervention using Acceptance and Commitment Therapy (ACT) technique to target and reduce emotional eating. The intervention will be modeled after Frayn and Knäuper's (2016) brief emotional eating intervention, which was derived from Forman et al.'s (2013) "Mind Your Health program". During the workshop, the following topics will be discussed, based on the three processes of ACT: (1) values clarification/commitment, (2) acceptance/distress tolerance, and (3) mindfulness/awareness.

SUMMARY:
Emotional eating is a behaviour that has been linked to weight concerns, mental health concerns, and disordered eating. Effective interventions have been developed to treat emotional eating, however these exist solely in the context of promoting weight loss. Emotional eating is not exclusive to those who struggle with weight and thus interventions are needed that target those who engage in emotional eating regardless of their weight status. The present study aims to do so through the implementation of a one day Acceptance and Commitment Therapy (ACT) workshop for emotional eaters.

DETAILED DESCRIPTION:
Emotional eating is defined as increased food consumption in response to negative emotions, and has been linked to weight concerns, mental health concerns, and disordered eating behaviours. Effective interventions have been developed that address emotional eating, namely to improve weight loss. Such interventions are based in Acceptance and Commitment Therapy (ACT), which encourages tolerance of internal cues, such as emotions, and external cues, such as food.

Emotional eating, however, is not exclusive to those who struggle with their weight. Many individuals maintain a normal weight despite engaging in emotional eating. These individuals still consume an excess of high calorie (for which they somehow eventually compensate), high fat, and high sugar foods as part of their emotional eating. Unhealthy dietary habits such as these have been shown to be associated with an increased risk of all-cause mortality, as well as health concerns including diabetes and cardiovascular disease. Individuals with normal weight are not eligible for ACT programs described above, despite the increased risk of health concerns associated with emotional eating.

The present study aims to test the feasibility and acceptability of a one-day ACT workshop to reduce emotional eating and improve health that is not focused on weight loss as its primary outcome, and rather targets all individuals who engage in emotional eating.

ELIGIBILITY:
Inclusion Criteria:

* Engaging in emotional eating as per a DEBQ-EE score of 3.25 or higher
* Being over the age of 18

Exclusion Criteria:

* Not meeting the DEBQ-EE 3.25 or higher inclusion criteria
* Being under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Intervention is open to all participants regardless of gender identity.
Enrollment: 32 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-03-05 (Actual); Study Completion 2019-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mallory Frayn, PhD (c), Principal Investigator — McGill University; Bärbel Knäuper, PhD, Principal Investigator — McGill University
Locations (1):
- McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Study data, including the intervention manual, study protocol, statistical analysis plan, and outcomes will be shared with other researchers upon request.
Supporting Information: Study Protocol, SAP
Time Frame: Upon publication of the study results.
Access Criteria: Upon request from other researchers.

REFERENCES:
- [Background] Forman EM, Butryn ML, Juarascio AS, Bradley LE, Lowe MR, Herbert JD, Shaw JA. The mind your health project: a randomized controlled trial of an innovative behavioral treatment for obesity. Obesity (Silver Spring). 2013 Jun;21(6):1119-26. doi: 10.1002/oby.20169. Epub 2013 May 13. PMID 23666772
- [Background] Geliebter A, Aversa A. Emotional eating in overweight, normal weight, and underweight individuals. Eat Behav. 2003 Jan;3(4):341-7. doi: 10.1016/s1471-0153(02)00100-9. PMID 15000995
- [Background] Hou L, Li F, Wang Y, Ou Z, Xu D, Tan W, Dai M. Association between dietary patterns and coronary heart disease: a meta-analysis of prospective cohort studies. Int J Clin Exp Med. 2015 Jan 15;8(1):781-90. eCollection 2015. PMID 25785058
- [Background] Konttinen H, Mannisto S, Sarlio-Lahteenkorva S, Silventoinen K, Haukkala A. Emotional eating, depressive symptoms and self-reported food consumption. A population-based study. Appetite. 2010 Jun;54(3):473-9. doi: 10.1016/j.appet.2010.01.014. Epub 2010 Feb 4. PMID 20138944
- [Background] Lillis J, Niemeier HM, Thomas JG, Unick J, Ross KM, Leahey TM, Kendra KE, Dorfman L, Wing RR. A randomized trial of an acceptance-based behavioral intervention for weight loss in people with high internal disinhibition. Obesity (Silver Spring). 2016 Dec;24(12):2509-2514. doi: 10.1002/oby.21680. Epub 2016 Nov 2. PMID 27804255
- [Background] Oliver G, Wardle J, Gibson EL. Stress and food choice: a laboratory study. Psychosom Med. 2000 Nov-Dec;62(6):853-65. doi: 10.1097/00006842-200011000-00016. PMID 11139006
- [Background] Schwingshackl L, Schwedhelm C, Hoffmann G, Lampousi AM, Knuppel S, Iqbal K, Bechthold A, Schlesinger S, Boeing H. Food groups and risk of all-cause mortality: a systematic review and meta-analysis of prospective studies. Am J Clin Nutr. 2017 Jun;105(6):1462-1473. doi: 10.3945/ajcn.117.153148. Epub 2017 Apr 26. PMID 28446499
- [Background] Sami W, Ansari T, Butt NS, Hamid MRA. Effect of diet on type 2 diabetes mellitus: A review. Int J Health Sci (Qassim). 2017 Apr-Jun;11(2):65-71. PMID 28539866
- [Background] van Strien T, van de Laar FA, van Leeuwe JF, Lucassen PL, van den Hoogen HJ, Rutten GE, van Weel C. The dieting dilemma in patients with newly diagnosed type 2 diabetes: does dietary restraint predict weight gain 4 years after diagnosis? Health Psychol. 2007 Jan;26(1):105-12. doi: 10.1037/0278-6133.26.1.105. PMID 17209703
- [Derived] Frayn M, Khanyari S, Knauper B. A 1-day acceptance and commitment therapy workshop leads to reductions in emotional eating in adults. Eat Weight Disord. 2020 Oct;25(5):1399-1411. doi: 10.1007/s40519-019-00778-6. Epub 2019 Sep 20. PMID 31541426

RESULTS

PARTICIPANT FLOW:
Groups:
- ACT Workshop for Emotional Eating: All participants were assigned to an ACT workshop designed to reduce emotional eating through the teaching of three skills: (1) values clarification/commitment, (2) acceptance/distress tolerance, and (3) mindfulness.
Period: Overall Study
Arm/Group | ACT Workshop for Emotional Eating
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ACT Workshop for Emotional Eating
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.71 (13.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnic group: Caucasian | 25
  Ethnic group: Middle Eastern | 1
  Ethnic group: Black | 1
  Ethnic group: Hispanic | 1
  Ethnic group: Other | 4
Region of Enrollment [Number; unit: participants]
  Canada | 32
Dutching Eating Behavior Questionnaire-emotional eating [Mean (Standard Deviation); unit: units on a scale] — Emotional eating, as assessed by the Dutch Eating Behaviour Questionnaire Emotional Eating Subscale (DEBQ-EE). Participants are asked to rate the frequency with which they engage in particular eating behaviours, on a 5-point Likert-type rating scale from never (1) to very often (5), with higher scores reflecting higher emotional eating. Only the emotional eating subscale of the DEBQ will be assessed and is calculated by averaging the 13 items that assess emotional eating.
  units on a scale | 3.91 (0.46)
Distress Tolerance Scale [Mean (Standard Deviation); unit: units on a scale] — Distress tolerance, as assessed by the Distress Tolerance Scale (DTS). Participants are asked to indicate the extent to which they agree with statements aimed at assessing distress tolerance, absorption, appraisal, and regulation from 1 (strongly agree) to 5 (strongly disagree), with lower scores reflecting lower distress tolerance. Subscale scores are derived by calculating the means of the items that make up each subscale. Total score is calculating by averaging the four subscales.
  units on a scale | 3.32 (0.92)
Food Craving Acceptance and Action Questionnaire [Mean (Standard Deviation); unit: units on a scale] — Food craving acceptance and action, as assessed by the Food Craving Acceptance and Action Questionnaire (FAAQ). Items are rated on a 6-point Likert-type rating scale from 1 (very seldom true) to 6 (always true), with higher scores reflecting higher acceptance. Total score is derived by summing all items.
  units on a scale | 28.18 (6.24)
Mindful Eating Questionnaire [Mean (Standard Deviation); unit: units on a scale] — Mindful eating, as assessed by the Mindful Eating Questionnaire (MEQ). It is a 28-item self-report measure that assesses five domains of mindful eating: disinhibition, external cues, awareness, emotional response and distraction. Participants are asked to indicate the extent to which extent they agree with each item from 1 ("never" / "rarely") to 4 ("usually"/ "always"), with higher scores reflecting higher levels of mindful eating. Total score is derived by taking the mean of the five subscales.
  units on a scale | 2.35 (0.35)
ACT Values Application [Mean (Standard Deviation); unit: units on a scale] — Application of ACT values techniques taught during the workshop, as assessed by items developed by the study's authors. Participants were asked to rate the extent to which they agreed with a number of value-based statements on a scale from 1 (strongly disagree) to 5 (strongly agree). Values score was derived by taking the mean of the items, with higher scores reflecting greater value-consistent eating behaviors.
  units on a scale | 3.24 (0.66)
Emotional eating frequency [Mean (Standard Deviation); unit: times per week] — As assessed by a self-report item developed by the study's authors. Participants were asked to report the number of times they engaged in emotional eating in the past week, from 1 (1 time) to 7 (7 or more times).
  times per week | 4.64 (1.66)
Ability to stop emotional eating [Mean (Standard Deviation); unit: units on a scale] — As assessed by a single self-report item developed by the study's authors. Participants were asked to report the number of instances in which they began to engage in emotional eating and were able to stop themselves, on a scale from 1 (none of the time) to 5 (very often).
  units on a scale | 1.96 (0.88)

OUTCOME MEASURES:

1. Primary Outcome: Emotional Eating - 2-weeks Post-intervention
Description: Emotional eating, as assessed by the Dutch Eating Behaviour Questionnaire Emotional Eating Subscale (DEBQ-EE). Participants are asked to rate the frequency with which they engage in particular eating behaviours, on a 5-point Likert-type rating scale from never (1) to very often (5), with higher scores reflecting higher emotional eating. Only the emotional eating subscale of the DEBQ will be assessed and is calculated by averaging the 13 items that assess emotional eating.
Time Frame: Assessed from baseline to 2-weeks post-intervention and 3-months post-intervention
Population: Based on incomplete questionnaire data, 28/32 participants were included in the final analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ACT Workshop for Emotional Eating
Number analyzed (Participants) | 28
units on a scale | 3.27 (0.58)

2. Primary Outcome: Emotional Eating - 3-months Post-Intervention
Description: as for outcome 1
Time Frame: Assessed from baseline to 2-weeks post-intervention and 3-months post-intervention
Population: Based on incomplete questionnaire data, 28/32 participants were included in the final analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ACT Workshop for Emotional Eating
Number analyzed (Participants) | 28
units on a scale | 3.10 (0.55)

3. Secondary Outcome: Distress Tolerance - 2-weeks Post-Intervention
Description: Distress tolerance, as assessed by the Distress Tolerance Scale (DTS). Participants are asked to indicate the extent to which they agree with statements aimed at assessing distress tolerance, absorption, appraisal, and regulation from 1 (strongly agree) to 5 (strongly disagree), with lower scores reflecting lower distress tolerance. Subscale scores are derived by calculating the means of the items that make up each subscale. Total score is calculating by averaging the four subscales.
Time Frame: Assessed from baseline to 2-weeks post-intervention and 3-months post-intervention
Population: Based on incomplete questionnaire data, 28/32 participants were included in the final analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ACT Workshop for Emotional Eating
Number analyzed (Participants) | 28
units on a scale | 3.17 (0.79)

4. Secondary Outcome: Distress Tolerance - 3-months Post-Intervention
Description: as for outcome 3
Time Frame: Assessed from baseline to 2-weeks post-intervention and 3-months post-intervention
Population: Based on incomplete questionnaire data, 28/32 participants were included in the final analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ACT Workshop for Emotional Eating
Number analyzed (Participants) | 28
units on a scale | 2.87 (0.86)

5. Secondary Outcome: Food Craving Acceptance and Action - 2-weeks Post-intervention
Description: Food craving acceptance and action, as assessed by the Food Craving Acceptance and Action Questionnaire (FAAQ). Items are rated on a 6-point Likert-type rating scale from 1 (very seldom true) to 6 (always true), with higher scores reflecting higher acceptance. Total score is derived by summing all items. Minimum score is 10 and maximum score is 60.
Time Frame: Assessed from baseline to 2-weeks post-intervention and 3-months post-intervention
Population: Based on incomplete questionnaire data, 28/32 participants were included in the final analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ACT Workshop for Emotional Eating
Number analyzed (Participants) | 28
units on a scale | 32.71 (4.29)

6. Secondary Outcome: Food Craving Acceptance and Action - 3-months Post-intervention
Description: as for outcome 5
Time Frame: Assessed from baseline to 2-weeks post-intervention and 3-months post-intervention
Population: Based on incomplete questionnaire data, 28/32 participants were included in the final analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ACT Workshop for Emotional Eating
Number analyzed (Participants) | 28
units on a scale | 32.68 (4.76)

7. Secondary Outcome: Mindful Eating - 2-weeks Post-intervention
Description: Mindful eating, as assessed by the Mindful Eating Questionnaire (MEQ). It is a 28-item self-report measure that assesses five domains of mindful eating: disinhibition, external cues, awareness, emotional response and distraction. Participants are asked to indicate the extent to which extent they agree with each item from 1 ("never" / "rarely") to 4 ("usually"/ "always"), with higher scores reflecting higher levels of mindful eating. Total score is derived by taking the mean of the five subscales.
Time Frame: Assessed from baseline to 2-weeks post-intervention and 3-months post-intervention
Population: Based on incomplete questionnaire data, 28/32 participants were included in the final analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ACT Workshop for Emotional Eating
Number analyzed (Participants) | 28
units on a scale | 2.51 (0.35)

8. Secondary Outcome: Mindful Eating - 3-months Post-intervention
Description: as for outcome 7
Time Frame: Assessed from baseline to 2-weeks post-intervention and 3-months post-intervention
Population: Based on incomplete questionnaire data, 28/32 participants were included in the final analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ACT Workshop for Emotional Eating
Number analyzed (Participants) | 28
units on a scale | 2.65 (0.41)

9. Secondary Outcome: ACT Values Application - 2-weeks Post-intervention
Description: Application of ACT values techniques taught during the workshop, as assessed by items developed by the study's authors. Participants were asked to rate the extent to which they agreed with a number of value-based statements on a scale from 1 (strongly disagree) to 5 (strongly agree). Values score was derived by taking the mean of the items, with higher scores reflecting greater value-consistent eating behaviors.
Time Frame: Assessed from baseline to 2-weeks post-intervention and 3-months post-intervention
Population: Based on incomplete questionnaire data, 28/32 participants were included in the final analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ACT Workshop for Emotional Eating
Number analyzed (Participants) | 28
units on a scale | 3.79 (0.63)

10. Secondary Outcome: ACT Values Application - 3-months Post-intervention
Description: as for outcome 9
Time Frame: Assessed from baseline to 2-weeks post-intervention and 3-months post-intervention
Population: Based on incomplete questionnaire data, 28/32 participants were included in the final analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ACT Workshop for Emotional Eating
Number analyzed (Participants) | 28
units on a scale | 3.63 (0.66)

11. Secondary Outcome: Emotional Eating Frequency - 2-weeks Post-intervention
Description: As assessed by a self-report item developed by the study's authors. Participants were asked to report the number of times they engaged in emotional eating in the past week.
Time Frame: Assessed from baseline to 2-weeks post-intervention and 3-months post-intervention
Population: Based on incomplete questionnaire data, 28/32 participants were included in the final analyses.
Measure: Mean (Standard Deviation); unit: times per week
Arm/Group | ACT Workshop for Emotional Eating
Number analyzed (Participants) | 28
times per week | 3.00 (1.49)

12. Secondary Outcome: Emotional Eating Frequency - 3-months Post-intervention
Description: as for outcome 11
Time Frame: Assessed from baseline to 2-weeks post-intervention and 3-months post-intervention
Population: Based on incomplete questionnaire data, 28/32 participants were included in the final analyses.
Measure: Mean (Standard Deviation); unit: times per week
Arm/Group | ACT Workshop for Emotional Eating
Number analyzed (Participants) | 28
times per week | 3.43 (1.67)

13. Secondary Outcome: Ability to Stop Emotional Eating - 2-weeks Post-intervention
Description: As assessed by a single self-report item developed by the study's authors. Participants were asked to report the number of instances in which they began to engage in emotional eating and were able to stop themselves, on a scale from 1 (none of the time) to 5 (very often).
Time Frame: Assessed from baseline to 2-weeks post-intervention and 3-months post-intervention
Population: Based on incomplete questionnaire data, 28/32 participants were included in the final analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ACT Workshop for Emotional Eating
Number analyzed (Participants) | 28
units on a scale | 2.68 (1.12)

14. Secondary Outcome: Ability to Stop Emotional Eating - 3-months Post-intervention
Description: as for outcome 13
Time Frame: Assessed from baseline to 2-weeks post-intervention and 3-months post-intervention
Population: Based on incomplete questionnaire data, 28/32 participants were included in the final analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ACT Workshop for Emotional Eating
Number analyzed (Participants) | 28
units on a scale | 2.71 (1.01)

15. Secondary Outcome: Feasibility Data: Recruitment, Eligibility, Attendance, and Attrition Rates
Description: These include recruitment, eligibility, attendance, and attrition rates
Time Frame: Assessed throughout the duration of the study from the recruitment period to the completion of the workshops and follow-up questionnaires (i.e., over a 3-month period).
Population: The population of analysis were the 59 individuals who initially expressed interest in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | ACT Workshop for Emotional Eating
Number analyzed (Participants) | 59
Participants
  Recruitment | 59
  Eligibility | 44
  Attendance | 32
  Attrition | 2

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the duration that each participant participated in the study (from baseline to 3-months post-intervention).
Arm/Group | ACT Workshop for Emotional Eating
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-09-16): https://cdn.clinicaltrials.gov/large-docs/80/NCT03744780/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-16): https://cdn.clinicaltrials.gov/large-docs/80/NCT03744780/SAP_001.pdf